CLINICAL TRIAL: NCT05918354
Title: Development and Evaluation of an Artificial Intelligence Model to Support Read Out of Skin Prick Automated Test Results for the Diagnosis of Aeroallergies
Brief Title: Development and Evaluation of an Artificial Intelligence Model for the Diagnosis of Aeroallergies
Acronym: SPAT_AI
Status: Completed | Type: Observational
Sponsor: Hippocreates (Industry)
Responsible Party: Sponsor
Other Study IDs: HDX003
Record Dates: First submitted 2023-06-15; First posted 2023-06-26 (Actual); Last update posted 2024-10-16 (Actual); Status verified 2024-10

CONDITIONS: Allergy
MeSH Terms: conditions — Hypersensitivity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Allergy: Adults aged 18 years or above, consulting the outpatient clinic for an allergy diagnosis to aeroallergens with skin prick automated test device.
  Interventions: Device: Skin Prick Automated Test

INTERVENTIONS:
Device: Skin Prick Automated Test — Detection of sensitisation to specific allergens via the skin prick automated test.

SUMMARY:
To improve accuracy and take out human error, Hippo Dx previously developed S.P.A.T., an automated skin prick test. Now, Hippo Dx will develop and evaluate a S.P.A.T. artificial intelligence (AI) medical software to support physicians in the read out of the test results from an automated skin prick test.

In this study 700 images will be collected to develop the AI model, an additional 200 images will be collected to evaluate performance of the AI model. In a last independent cohort of 100 patients, performance of read-out by the physician will be compared with read out by the physician supported by the S.P.A.T. AI medical software.

The primary endpoint is the accuracy of the maximal wheal size measurement by S.P.A.T. AI versus the maximal wheal size measurement by the physician.

It is a prospective multicentric study that will include 1000 study participants from different countries.

ELIGIBILITY:
Inclusion Criteria:

- Adults aged 18 years or above, consulting the outpatient clinic for an allergy diagnosis to aeroallergens will be included.

Exclusion Criteria:

* Skin pathology like chronic or exuberant urticaria, dermographism, chronic dermatitis that needs daily treatment
* Use of antihistaminic medication < 7 days before the start of the study
* Use of tricyclic antidepressants (antihistamine activity) < 7 days before the start of the study
* Use of topical corticoids on the forearm < 7 days before the start of the study
* Use of Omalizumab < 6 months before the start of the study
* Pregnancy: there is a remote possibility of inducing a systemic allergic reaction that could induce uterine contractions or necessitate the use of epinephrine (thought to cause constriction of the umbilical artery)
* Incapacitated individuals
* Individuals who do not speak the local language (Dutch - French)
* Individuals who cannot read or write

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults aged 18 years or above, consulting the outpatient clinic for an allergy diagnosis to aeroallergens will be included.
Sampling Method: Non-Probability Sample
Enrollment: 993 (Actual)
Dates: Start 2023-07-10 (Actual); Primary Completion 2024-09-11 (Actual); Study Completion 2024-09-11 (Actual)

PRIMARY OUTCOMES:
Equivalency of S.P.A.T. artificial intelligence versus physician | 15 minutes after the diagnostic test
  The equivalency of the maximal wheal diameter as measured by S.P.A.T. AI versus the maximal wheal diameter as assessed by the physician.

SECONDARY OUTCOMES:
Precision of S.P.A.T. artificial intelligence versus physician | 15 minutes after the diagnostic test
  Likelihood that the S.P.A.T. AI maximal wheal diameter measurement lays within the range of the maximal wheal size measurement of 3 independent physicians.
Intra-reader variability of S.P.A.T. read out by physicians | 15 minutes after the diagnostic test
  Variation in maximal wheal size diameter of the same image by 3 independent physicians.
Comparison of different methods (maximal wheal diameter) of read out by S.P.A.T. artificial intelligence versus physician | 15 minutes after the diagnostic test
  Accuracy of the maximal wheal diameter by S.P.A.T. AI versus the maximal wheal diameter measurement by the physician.
Comparison of S.P.A.T. artificial intelligence supporting the physician versus physician | 15 minutes after the diagnostic test
  Inter-reader variability of read out of S.P.A.T. results by the physician supported by the S.P.A.T. AI software versus the physician alone.
Time impact of S.P.A.T. artificial intelligence supporting the physician versus physician | 15 minutes after the diagnostic test
  Total time required to perform read out of S.P.A.T. results by the physician supported by the S.P.A.T. AI software versus the physician alone.
Comparison of different methods (mean - maximal wheal diameter) of read out by S.P.A.T. artificial intelligence versus physician | 15 minutes after the diagnostic test
  Accuracy of mean wheal diameter by S.P.A.T. AI versus the maximal wheal diameter measurement by the physician.
Comparison of different methods (wheal area - maximal wheal diameter) of read out by S.P.A.T. artificial intelligence versus physician | 15 minutes after the diagnostic test
  Accuracy of wheal area by S.P.A.T. AI versus the maximal wheal diameter measurement by the physician.
Comparison of different methods (HEP index - maximal wheal diameter) of read out by S.P.A.T. artificial intelligence versus physician | 15 minutes after the diagnostic test
  Accuracy of HEP-index measurement by S.P.A.T. AI versus the maximal wheal diameter measurement by the physician.

CONTACTS AND LOCATIONS:
Overall Officials: Mark Jorissen, MD, PhD, Principal Investigator — UZ Leuven
Locations (6):
- Belgium (5):
  - Clinique Universitaires Saint-Luc, Brussels
  - Ziekenhuis Oost Limburg, Genk
  - UZ Leuven, Leuven
  - CHU de Liège, Liège
  - GZA ziekenhuizen, Wilrijk
- Klinikum rechts der Isar, Munich, Germany

IPD SHARING:
Plan to Share IPD: Undecided